CLINICAL TRIAL: NCT06050564
Title: Therapeutic Recommendations Based on Clinical History and Video Documented PBS-Score, an International Cross-sectional Multicenter Study
Brief Title: Therapeutic Recommendations Based on Clinical History and Video Documented PBS-Score
Status: Completed | Type: Observational
Sponsor: Region Stockholm (Other Government)
Responsible Party: Principal Investigator, Eva Weidenhielm-Brostrom, Professor, Region Stockholm
Other Study IDs: K2022-10587
Record Dates: First submitted 2023-09-11; First posted 2023-09-22 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Clubfoot
Keywords: PBS-score; PEVA; Treatment clubfoot
MeSH Terms: conditions — Clubfoot

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Treatment recommendations will be based on video documented PBS-Score — Therapeutic recommendations from orthopedic surgeons, will be summarized and described

SUMMARY:
Determine the relationship between the PBS-score and treatment recommendations provided by senior pediatric orthopedic surgeons.

DETAILED DESCRIPTION:
In conjunction with the assessments of video documented PBS-score items (described in Study I), treatment recommendations from six to eight experienced pediatric orthopedic surgeons from four different countries will be collected. Their recommendations will be based on the included items of the PBS-score, and patient history including age of the child, Pirani score, initial treatment (need for tenotomy), and reported compliance to orthotic use.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of idiopathic clubfoot, ability to walk 10 m repeatedly, and ability to communicate verbally (and in writing for caregivers) in Swedish, English, Portuguese, Urdu, or Pashto.

Exclusion Criteria:

* syndromic clubfoot

Ages: 4 Years to 14 Years | Sex: All
Age Groups: Child
Study Population: 120 children with idiopathic clubfoot will be included from four different countries
Sampling Method: Non-Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2023-01-10 (Actual); Primary Completion 2023-12-28 (Actual); Study Completion 2024-06-18 (Actual)

PRIMARY OUTCOMES:
Treatment recommendations | 1 year
  Treatment recommendations from eight to ten experienced pediatric orthopedic surgeons will be collected. Their recommendations will be based on the included items of the Pirani Böhm Sinclair, PBS-score, the lowest score with 7 points being the best and 18 points the worst. The patient history including age of the child, Pirani score minimum 0 and maximum score is 6, the higher, the more severe deformity. Initial treatment (need for Achilles tenotomy), and reported compliance to orthotic use.

CONTACTS AND LOCATIONS:
Overall Officials: Eva W Broström, Professor, Principal Investigator — Astrid Lindgren Children´s Hospital
Locations (1):
- Astrid Lindgren Children´s Hospital, Stockholm, Region Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No